CLINICAL TRIAL: NCT03034668
Title: The Acute and Chronic Influence of a Botanical Supplement on Muscle Function and Lean Body Mass
Brief Title: Botanical Supplement Muscle Function and Lean Body Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Givaudan France Naturals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 16-1991
Record Dates: First submitted 2017-01-17; First posted 2017-01-27 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteers
Keywords: Botanical Supplement; Performance-Enhancing Supplement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CS16-003 Full dose (Experimental): 350 mg capsule QD Rhodiola rosea L. & Rhaptonticum carthamoides extracts
  Interventions: Dietary Supplement: CS16-003 Full dose
- CS16-003 Half dose (Experimental): 175 mg capsule QD 50% Rhodiola rosea L. & Rhaptonticum carthamoides extracts + 50% Maltodextrin
  Interventions: Dietary Supplement: CS16-003 Half dose
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CS16-003 Full dose — 350 mg 'Rhodiola rosea L. & Rhaptonticum carthamoides extracts
  Arms: CS16-003 Full dose
Dietary Supplement: CS16-003 Half dose — 175 mg 'Rhodiola rosea L. & Rhaptonticum carthamoides extracts + maltodextrin 175 mg
  Arms: CS16-003 Half dose
Dietary Supplement: Placebo — Maltodextrin: 350 mg
  Arms: Placebo

SUMMARY:
Purpose: To evaluate the acute and chronic effects of a botanical supplement on strength, muscle function, and lean body mass

Participants: The acute phase will include 30 participants, and the chronic phase will include 84 participants. All participants must be healthy recreationally active males between the ages of 18 and 35 years.

Procedures (methods):

Acute phase: Participants will complete three testing visits as part of as part of a cross-over design, during which strength and muscle function will be assessed prior to and following consumption of a supplement. The experimental supplement is a blend of the botanical extracts; treatment arms will include a full dose (FULL; 350 mg capsule), half dose (HALF; 175 mg plus maltodextrin), or placebo (PLA; maltodextrin).

Chronic phase: Body composition, muscle cross-sectional area, a complete blood count and metabolic panel, subjective surveys, and strength will be measured prior to and following an 8-week supervised resistance training program, in conjunction with daily supplementation of FULL, HALF, or PLA.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally Active (1- 4 hours of exercise/ sports participation per week and no more than 1 hour of resistance training exercise per week) for the previous 12 weeks.
* BMI < 30 kg/m²
* Have not smoked in the past year.
* Participant has provided written and dated informed consent to participate in the study
* Participant is willing and able to comply with the protocol
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire
* Participant agrees to abstain from caffeine, tobacco, alcohol, and exercise within 24 hours of testing visits

Exclusion Criteria:

* Participant has not used any dietary supplements within 12 weeks prior to enrollment and will not begin supplementation during the study. Potential supplements include but are not limited to Beta-alanine, Creatine, HMB, Carnosine, Taurine, androstenedione, DHEA, Whey protein, or a pre-workout supplement.
* Participant has gained or lost 10 lbs in the previous 2 months.
* Participant is currently enrolled in a separate clinical trial.
* Participant has participated in a clinical trial within the previous 2 months that includes modifications to their physical and/or diet.
* Participant has a known allergy or sensitivity to the placebo (maltodextrin) or active ingredients (Rhodiola & Rhaptonicum)
* Participant consumes more than 8 cups (1 cup = 6 oz) of coffee per day on a regular basis
* Participant consumes more than 3 alcoholic drinks per day.
* Participant uses recreational drugs daily.
* Previous physical symptoms causing a physician to recommend you to refrain from exercise.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2016-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Maximal Isokinetic Leg Extension strength measured by dynamometry | Acute/Immediate
Maximal Upper and Lower Body Strength measured by 1 repetition maximum | 8 weeks

SECONDARY OUTCOMES:
Bench Press Repetitions to Fatigue | 8 weeks
Leg Press Repetitions to Fatigue | 8 weeks
Body Composition-Lean Mass | 8 weeks
Body Composition-Fat Mass | 8 weeks
Muscle cross sectional area | 8 weeks
Change in Quality of Life Score from baseline to 8 weeks | baseline, 8 weeks
  Quality of life from a visual analog scale (VAS) 0-100, with 0 = worst quality of life and 100=best quality of life.
Change in Felt Arousal score from baseline to 8 weeks | baseline, 8 weeks
  Felt arousal scale. Scores range 1-6 with 1 being low arousal and 6 being high. One score selected.
Change in Mood score from baseline to 8 weeks | baseline; 8 weeks
  Mood determined from a VAS. 0-100, with 0 = not depressed at all and 100 = most depressed.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Department of Exercise and Sport Science, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No